CLINICAL TRIAL: NCT07264764
Title: Evaluation of Optic Nerve Sheath Diameter, Cerebral Oxygen Saturation and Cognitive Functions in Patients Undergoing Laparoscopic Abdominal Surgeries; Prospective Observational Study
Brief Title: Optic Nerve Sheath Diameter and Postoperative Cognitive Disfunction at Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, gulbin sezen, professor, Duzce University
Other Study IDs: DuzceU-GYSezen-005
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: optic nerve sheath diameter; laparoscopic surgery; postoperative cognitive dysfunction; regional cerebral oxygen saturation
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- laparoscopic abdominal surgery: Fifty adult patients (aged 20-60 years; ASA I-III) scheduled for elective laparoscopic abdominal surgery (e.g., cholecystectomy, appendectomy, hernia repair) under general anesthe-sia were enrolled. All patients underwent standardized anesthetic management. Following preoxygenation with 100% oxygen for 2 minutes, anesthesia induction consisted of intravenous thiopental sodium (5-7 mg·kg-¹), fentanyl (1 µg·kg-¹), rocuronium (0.6 mg·kg-¹), and lidocaine (1 mg·kg-¹). Tracheal intubation was performed by an experienced anesthesiologist, with laryngoscopy duration recorded. Anesthesia was maintained with 1 minimum alveolar concentration (MAC) sevoflurane in 50% O2/air mixture, using volume-controlled ventilation (tidal volume 6-8 mL·kg-¹, PEEP 5 cmHO2, respiratory rate adjusted to maintain end-tidal CO2 [EtCO2] 33-40 mmHg). Hemodynamic variables, and peak inspiratory airway pressure (Ppeak) were continuously recorded.
  Interventions: Diagnostic Test: Optic nerve sheath diameter (ONSD)

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter (ONSD) — All parameters (ONSD, rSO2, IAP, EtCO2, Ppeak, SBP, DBP, MAP, HR) were recorded at:T0: Pre-induction baseline,T1: 5 min after induction,T2: 5 min after COpneumoperitoneum,T3: 30 min after pneumoperitoneum,T4: 5 min post-desufflation. ONSD was measured using a high-frequency (18 MHz) linear ultrasound probe (Mylab 5, Esaote, Genoa, Italy). The ONSD was defined as the distance between the outer edges of the optic nerve sheath 3 mm posterior to the optic disc. rSO2 was measured continuously using NIRS (INVOS 4100) with bilateral frontal sensors. MMSE, administered in a face-to-face format by a trained researcher on the day before surgery (baseline) and 24 hours postoperatively. A decline of ≥2 points in the postoperative score compared to baseline was considered indicative of postoperative cognitive dysfunction (POCD).

SUMMARY:
Purpose:

Pneumoperitoneum during laparoscopic abdominal surgery increases intra-abdominal pressure (IAP), potentially altering intracranial pressure (ICP) and cerebral oxygenation, with unclear implications for early postoperative cognitive dysfunction (POCD). Optic nerve sheath diameter (ONSD) via ultrasonography and near-infrared spectroscopy (NIRS) based cerebral oximetry offer non-invasive monitoring tools to assess these changes.

DETAILED DESCRIPTION:
In this prospective observational study, fifty ASA I-III patients (20-60 years) undergoing elective laparoscopic abdominal surgery under general anesthesia were enrolled. Serial measurements of bilateral ONSD and regional cerebral oxygen saturation (rSO2, NIRS) were obtained at five perioperative time points: before induction (T0), 5 minutes post-induction (T1), 5 minutes after CO2 pneumoperitoneum (T2), 30 minutes after pneumoperitoneum (T3), and 5 minutes post-desufflation (T4). IAP was measured both intravesically and via insufflator readings. Cognitive function was assessed using the Mini-Mental State Examination (MMSE) preoperatively and at 24 hours postoperatively. Hemodynamic parameters and airway pressures were recorded concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years;
* American Society of Anesthesiologists [ASA] I-III)
* scheduled for elective laparoscopic abdominal surgery (e.g., cholecystectomy, appendectomy, hernia repair) under general anesthesia

Exclusion Criteria:

* pregnancy,
* known neurological or ocular disease,
* prior ocular surgery,
* significant cardiovascular disease (moderate to severe),
* chronic obstructive pulmonary disease (COPD),
* conversion from laparoscopy to open laparo-tomy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Aged 20-60 years, ASA I-III, all patients who will undergo upper abdominal surgery without any excluded criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) | • T0: Pre-induction baseline • T1: 5 minutes after induction • T2: 5 minutes after CO pneumoperitoneum • T3: 30 minutes after pneumoperitoneum • T4: 5 minutes post-desufflation
  ONSD was measured by a single trained anesthesiologist using a high-frequency (18 MHz) linear ultrasound probe (Mylab 5, Esaote, Genoa, Italy). With patients in the supine position and eyelids closed, the probe was gently placed on the upper eyelid in horizontal and vertical planes without exerting pressure. The ONSD was defined as the distance between the outer edges of the optic nerve sheath 3 mm posterior to the optic disc.

SECONDARY OUTCOMES:
postoperative cognitive dysfunction | Time 1: Preoperative one day before Time 2: Postoperative 24 hours
  Cognitive performance was evaluated using the Mini-Mental State Examination (MMSE), administered in a face-to-face format by a trained researcher on the day before surgery (baseline) and 24 hours postoperatively.The Mini Mental State Examination (MMSE) test consists of 11 questions and is evaluated from a minimum score of 0 to a maximum of 30, below 24 point is considered worse outcome, while a decline of ≥2 points in the postoperative score compared to baseline was considered indicative of postoperative cognitive dysfunction (POCD), consistent with prior studies.
cerebral oxygenation | T0: Pre-induction baseline • T1: 5 minutes after induction • T2: 5 minutes after CO pneumoperitoneum • T3: 30 minutes after pneumoperitoneum • T4: 5 minutes post-desufflation
  Regional cerebral oxygen saturation (rSO2) was measured continuously using near-infrared spectroscopy (NIRS; INVOS 4100, Medtronic, Minneapolis, MN, USA) with bilateral frontal sensors.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Medicine School, Anesthesiology and Reanimation Department, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou J, Li J, Ye T, Zeng Y. Ultrasound measurements versus invasive intracranial pressure measurement method in patients with brain injury: a retrospective study. BMC Med Imaging. 2019 Jul 5;19(1):53. doi: 10.1186/s12880-019-0354-0. PMID 31277606
- [Background] Amini A, Kariman H, Arhami Dolatabadi A, Hatamabadi HR, Derakhshanfar H, Mansouri B, Safari S, Eqtesadi R. Use of the sonographic diameter of optic nerve sheath to estimate intracranial pressure. Am J Emerg Med. 2013 Jan;31(1):236-9. doi: 10.1016/j.ajem.2012.06.025. Epub 2012 Aug 31. PMID 22944553
- [Background] Demirgan S, Ozcan FG, Gemici EK, Guneyli HC, Yavuz E, Gulcicek OB, Selcan A. Reverse Trendelenburg position applied prior to pneumoperitoneum prevents excessive increase in optic nerve sheath diameter in laparoscopic cholecystectomy: randomized controlled trial. J Clin Monit Comput. 2021 Feb;35(1):89-99. doi: 10.1007/s10877-020-00608-6. Epub 2020 Oct 21. PMID 33089454
- [Result] Jo YY, Kim JY, Lee MG, Lee SG, Kwak HJ. Changes in cerebral oxygen saturation and early postoperative cognitive function after laparoscopic gastrectomy: a comparison with conventional open surgery. Korean J Anesthesiol. 2016 Feb;69(1):44-50. doi: 10.4097/kjae.2016.69.1.44. Epub 2016 Jan 28. PMID 26885301
- [Result] Keller DS, Senagore AJ, Fitch K, Bochner A, Haas EM. A new perspective on the value of minimally invasive colorectal surgery-payer, provider, and patient benefits. Surg Endosc. 2017 Jul;31(7):2846-2853. doi: 10.1007/s00464-016-5295-x. Epub 2016 Nov 4. PMID 27815745